CLINICAL TRIAL: NCT05282784
Title: Exploratory, Open-labelled, Control Group-included, Single Institution Clinical Trial for Evaluating Immunogenic Effect of Hyperthermia Applied With Flexible Electrode-typed 2-MHz Device During Radiotherapy for Solid Tumors
Brief Title: Hyperthermia With Flexible Electrode-typed 2-MHz Device During Radiotherapy for Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei Hyperthermia Study Group (Other)
Collaborators: Medicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YURO-H8
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor
Keywords: Radiotherapy; Hyperthermia
MeSH Terms: conditions — Hyperthermia | interventions — Diathermy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermia group (Experimental): Hyperthermia Radiotherapy
  Interventions: Other: Hyperthermia; Radiation: Radiotherapy
- Control (Active Comparator): Radiotherapy
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Other: Hyperthermia — Patients will be treated with hyperthermia 2 or 3 times a week. Treatment will be performed for 1 hours per each visit.
  Patients will be treated with radiotherapy 5 times a week.
  Arms: Hyperthermia group
Radiation: Radiotherapy — Patients will be treated with radiotherapy 5 times a week.

SUMMARY:
The main purpose of this study is to evaluate immunogenic effect of hyperthermia applied with flexible electrode-typed 2-MHz device during radiotherapy for solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor (primary, metastatic)
* Eastern Cooperative Oncology Group (ECOG) score 0-3
* Ability to understand and the willingness to sign a written informed consent documents

Exclusion Criteria:

* Myocardial infarct, unstable angina, heart failure, uncontrolled arrhythmia within 6 months
* Active infectious disease
* Pregnant or probability of pregnancy during treatment
* Obesity (BMI ≥35)
* Immunosuppressive drug after organ transplantation
* Autoimmune disease
* Skin injury on treatment area

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenic effect | 1 weeks after treatment
  NK cell, CD4+ T cell, CD8+ T cell